CLINICAL TRIAL: NCT02008851
Title: A Phase 1, Open-Label Safety and Tolerability Study of an Autologous Neo-Kidney Augment (NKA) in Patients With Type 2 Diabetes and Chronic Kidney Disease
Brief Title: A Phase 1, Open-label Safety Study of NKA in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Tengion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TNG-CL011
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Type 2 Diabetes; Neo-kidney augment; Regenerative medicine
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantation of Neo-kidney Augment (Experimental): Patients receiving one dose (implant) of NKA into the left kidney
  Interventions: Biological: Neo-kidney augment

INTERVENTIONS:
Biological: Neo-kidney augment — Injection of 3.0 x 10e6 selected renal cells into the left kidney of the patient

SUMMARY:
The purpose of this study is to determine if selected renal cells, obtained by biopsy from a patient with chronic kidney disease (CKD) and Type 2 Diabetes (i.e., autologous cells) can be safely implanted back into the patient.

DETAILED DESCRIPTION:
This is a Phase 1 safety and tolerability study to determine if NKA, manufactured from a patient's renal biopsy tissue, can be safely implanted back into the kidney of the patient. Patients must have CKD and Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus (T2DM).
* Patients with CKD defined as glomerular filtration rate (GFR) of 20 - 50 mL/min/1.73m2, inclusive.
* Microalbuminuria that cannot be explained by an alternative diagnosis. Microalbuminuria is defined as a urinary albumin-creatinine ration (UACR) ≥ 30 mg/g or urine albumin excretion ≥ 30 mg/day on 24 hour urine collection.
* Ongoing treatment with ACEi or ARB. Patients who are intolerant may be included as long as they have stable blood pressure.
* Systolic blood pressure between 105 and 140 mmHg (inclusive) and diastolic blood pressure ≤ 90 mmHg.
* The patient should have historical data to provide a reasonable estimate of the rate of progression of CKD

Exclusion Criteria:

* Type 1 diabetes mellitus (DM).
* History of a renal transplant.
* HbA1c > 10% at Screening.
* Hemoglobin levels < 9 g/dL prior to biopsy or implant.
* Known allergy to kanamycin or structurally similar aminoglycoside antibiotics.
* Abnormal coagulation status as measured by activated partial prothrombin time, international normalized ratio (INR), and/or platelet count.
* Ineligible for a biopsy (e.g., based on size or cortical depth), MRI or renal scintigraphy study (e.g. due to hypersensitivity or allergy) according to standard site practices.
* Not a good candidate for laparoscopic surgical procedure (based on the assessment of the surgeon who will be performing the implant), including patients who are morbidly obese, have excessive fat surrounding the kidney, have a BMI > 45, or who are otherwise at excessive risk for serious complications.
* Clinically significant infection requiring parenteral antibiotics within 6 weeks of biopsy or implantation.
* Patients with small kidneys (average size < 9 cm) or only one kidney. Patients with a rapid decline in renal function over the last 3 months prior to biopsy or acute kidney injury.
* Patients with any of the following conditions prior to biopsy: renal tumors, polycystic kidney disease, renal cysts or other anatomic abnormalities that would interfere with the biopsy or implantation procedure (e.g., cysts in the pathway of the injection for implantation), hydronephrosis, skin infection over proposed biopsy sites, or evidence of a urinary tract infection.
* Female subjects who are pregnant, lactating (breast feeding) or planning a pregnancy during the course of the study.
* History of cancer within the past 3 years (excluding non-melanoma skin cancer and carcinoma in situ of the cervix).
* Life expectancy of less than 2 years.
* Any contraindication or known anaphylactic or severe systemic reaction to either human blood products or materials of animal (bovine, porcine) origin or anesthetic agents.
* Positive for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) assessed.
* Subjects with active tuberculosis (TB) requiring treatment in the past 3 years.
* Immunocompromised subjects or patients receiving immunosuppressive agents.
* Subjects with uncontrolled diabetes, incapacitating cardiac and/or pulmonary disorders.
* History of active alcohol and/or drug abuse that in the investigator's assessment would impair the subject's ability to comply with the protocol.
* Patients with clinically significant hepatic disease.
* Patients with bleeding disorders that would, in the opinion of the Investigator, interfere with the performance of study procedures; patients taking Coumarins (e.g.,Warfarin) or other anticoagulants (e.g. enoxaparin or direct thrombin inhibitors).
* Use of any investigational product within 3 months of the biopsy .

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events related to study procedures or investigational product | 12 months

SECONDARY OUTCOMES:
Number of renal-specific adverse events | 12 months

OTHER OUTCOMES:
Changes in renal function over time | 12 months
  Exploratory objectives include assessment of renal function over time; e.g., glomerular filtration rate (GFR), serum creatinine, and proteinuria.

CONTACTS AND LOCATIONS:
Overall Officials: Eric McAllister, MD, DPhil, Study Director — Tengion, Inc.
Locations (5):
- United States (5):
  - University of Chicago Medicine, Chicago, Illinois
  - LSU Health Care Services, New Orleans, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - UNC Medical Center, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee